CLINICAL TRIAL: NCT02758067
Title: Interventional, Randomised, Double-blind, Parallel-group, Active-comparator, Flexible-dose Study to Compare the Effectiveness of Brexpiprazole to That of Risperidone in Adult Patients With Schizophrenia
Brief Title: Comparison of the Effectiveness of Brexpiprazole With That of Risperidone
Acronym: TAILWIND
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was withdrawn for administrative reasons. There were no safety concerns.
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16758A; 2015-001749-97 (EudraCT Number)
Record Dates: First submitted 2016-04-29; First posted 2016-05-02 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — brexpiprazole; Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- brexpiprazole (Experimental)
  Interventions: Drug: brexpiprazole
- risperidone (Experimental)
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: brexpiprazole — 2- 4 mg/day, tablets, oral, 28-weeks
  Other Names: Rexulti (R)
  Arms: brexpiprazole
Drug: risperidone — 4-6 mg/day, tablets, oral, 28-weeks
  Arms: risperidone

SUMMARY:
To demonstrate that the effectiveness of brexpiprazole (2-4 mg/day) on quality of life is non-inferior to that of risperidone (4-6 mg/day) in adult patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* The patient has schizophrenia diagnosed according to DSM-5™
* The patient has his or her first formal diagnosis of schizophrenia less than 10 years ago
* The patient has been prescribed outpatient oral antipsychotic treatment at recommended dose range as stated in the Summary of product characteristics or equivalent document/label for the full 3 months prior to the Screening Visit.
* The patient has CGI-S score of 3 (mildly ill) or 4 (moderately ill) at the Screening and Baseline Visits.
* The patient has a Global Assessment Scale (GAS) score of 41 to 70 (limits included) at the Screening and Baseline Visits.
* The patient is in need of a change in the current antipsychotic treatment due to insufficient functional improvement and, in the judgement of the investigator, would benefit from a switch to another treatment. Reasons for switching include but are not limited to the following reasons:

  1. lack of adequate response to his or her current antipsychotic medication,
  2. poor tolerability to his or her current antipsychotic medication,
  3. unwillingness of the patient to adhere to his or her current antipsychotic medication.

Exclusion Criteria:

* The patient has a psychiatric disorder (DSM-5™ criteria) other than schizophrenia established as the primary diagnosis.
* The patient is experiencing acute exacerbation of psychotic symptoms at the Screening Visit, between the Screening and Baseline Visits or at the Baseline Visit.
* The patient is hospitalised for his or her psychotic symptoms at the Screening Visit, between the Screening and Baseline Visits or at the Baseline Visit.
* The patient is treated with brexpiprazole, risperidone or clozapine at the time of Screening Visit.
* The patient has shown, in the investigator's judgment, significant lack of efficacy to brexpiprazole, risperidone or paliperidone when treated at recommended dose range as stated in their respective Summary of product characteristics or equivalent document/ label, in a manner that would preclude benefiting from the study medication if randomised to brexpiprazole or risperidone during the study.
* The patient is considered resistant to antipsychotic treatment according to the investigator's judgement.
* The patient is at significant risk of harming himself/herself, or others according to the investigator's judgement or based on the Columbia Suicide Severity Rating Scale (C-SSRS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life (QLS total score) | Baseline to Week 28
  Evaluated by non-inferiority followed by superiority if non-inferiority is confirmed.
  The Quality of Life Scale (QLS) is a clinician-rated scale designed to assess deficit symptoms of schizophrenia and functioning during the preceding 4 weeks. The QLS consists of 21 items in 4 domains: Interpersonal Relations (eight items), Instrumental Role (four items), Intrapsychic Foundations (seven items), and Common Objects and Activities (two items). Each item is rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning). Definitions are provided for 4 anchor points of the 7 points. Each item has a brief description of the judgement to be made and a set of suggested probes for the clinician. The total score is calculated as the sum of all 21 items giving a range of 0 to 126, where the higher score indicates normal or unimpaired functioning

SECONDARY OUTCOMES:
Change in the 'Interpersonal Relations' QLS Domain Score | Baseline to Week 28
  The Interpersonal Relations domain score is the sum of 8 items (numbers 1 to 8). Each item is rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning), giving a range of 0 to 48, where the higher score indicates normal or unimpaired functioning
Change in the 'Instrumental Role' QLS Domain Score | Baseline to Week 28
  The Instrumental Role domain score is calculated as the sum of 4 items (numbers 9 to 12). Each item is rated on a 7-point scale, from 0 (severe where the higher score indicates normal or unimpaired functioning
Change in the 'Intrapsychic Foundations' QLS Domain Score | Baseline to Week 28
  The Intrapsychic Foundations domain score is calculated as the sum of 7 items (numbers 13 to 17 and 20 and 21). Each item is rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning), giving a range of 0 to 42, where the higher score indicates normal or unimpaired functioning
Change in the 'Common Objects and Activities' QLS Domain Score | Baseline to Week 28
  The Common Objects and Activities score is calculated as the sum of 2 items (numbers 18 and 19). Each item is rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning), giving a range of 0 to 12, where the higher score indicates normal or unimpaired functioning
Change in Global severity of illness (CGI-S) | Baseline to Week 28
  Clinical Global Impression - Severity of Illness (CGI-S) score provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients).
Investigator's Assessment Questionnaire (IAQ) Total Score | Baseline to Week 28
  The IAQ is a clinician-rated scale designed to assess the relative effectiveness (efficacy, safety and tolerability) of antipsychotic medications in patients with schizophrenia or schizoaffective disorder. The IAQ consists of 12 items: positive symptoms, negative symptoms, other efficacy symptoms, cognition, energy, mood, somnolence, weight gain, signs and symptoms of prolactin elevation, akathisia, extrapyramidal symptoms (EPS) (other than akathisia) and other safety or tolerability issues. For each item, the current medication is compared with previous antipsychotic medication on a five-point scale from 1 (Much better) to 5 (Much worse), or that item is Not applicable
Functional response (QLS total score) | at Week 28
  Defined as change from Baseline in QLS total score of ≥10 points
Readiness for Work Questionnaire (WoRQ) | Baseline to Week 28
  The Readiness for Work Questionnaire (WoRQ) is a clinician-rated scale designed to measure a schizophrenic patient's ability to work. The WoRQ total score is based on 7 statements. The statements is rated on a four-point scale, from 'strongly agree', 'agree', 'disagree' or 'strongly disagree'. Lower WoRQ total scores indicate better functioning
Work readiness status (from the WoRQ) | at Week 28
  The work readiness status is assessed by the clinician. The 7 statements from WoRQ are used to aid in reaching the dichotomous work readiness judgment where the clinician must indicate (yes or no) if the patient is ready for work or not
Time to discontinuation | from Baseline to Week 28

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com